CLINICAL TRIAL: NCT07027527
Title: A Phase 1b, Open-label, Randomized, Multicenter, Active Comparator Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of the Combination of APG777 + APG990 in Adults With Moderate-to-Severe Atopic Dermatitis
Brief Title: An Active Comparator Safety Study Evaluating the Combination of APG777 + APG990 in Moderate-to-Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Apogee Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG279-101
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Moderate-to-Severe AD; APG777; Dupilumab; APG990
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APG777 + APG990 (Experimental): Participants will receive protocol specified combination dose of APG777 + APG990
  Interventions: Drug: APG777; Drug: APG990
- Dupilumab (Active Comparator): Participants will receive protocol specified dose of Dupilumab
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: APG777 — Subcutaneous (SC) injection
  Arms: APG777 + APG990
Drug: APG990 — SC injection
  Arms: APG777 + APG990
Drug: Dupilumab — SC injection
  Other Names: Dupixent
  Arms: Dupilumab

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetic (PK) parameters of the combination of APG777 + APG990 in adults with moderate-to-severe atopic dermatitis (AD), in comparison to dupilumab. The duration of the study will be approximately 82 weeks for each participant and will consist of a Screening Period (up to 6 weeks), Treatment Period (Baseline-Week 24), and Follow-up Period (Week 28-Week 76).

DETAILED DESCRIPTION:
Participants will be randomized to APG777 + APG990 or dupilumab in a 1:1 ratio. Randomization will be stratified on Day 1 according to Baseline disease severity and geographic region.

ELIGIBILITY:
Inclusion Criteria

* Have a diagnosis of AD that has been present for ≥ 1 year prior to the Screening visit and as determined by the Investigator through participant interview and/or review of the medical history.
* Moderate-to-severe AD at Screening and Baseline (Day 1) visits, defined as: a) Eczema Area and Severity Index (EASI) score of ≥ 16, b) vIGA-AD score of ≥ 3, and c) AD affecting ≥10% of body surface area (BSA).
* History of inadequate response to treatment with topical medications
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 1) visit.

Exclusion Criteria

* Participation in a prior study with APG777 or APG990.
* Prior treatment with protocol-specified monoclonal antibodies (mAbs).
* Has used any AD-related topical medications within 7 days prior to Baseline visit.
* Has used systemic treatments (other than biologics) and/or phototherapies and/or laser therapy that could affect AD within 4 weeks prior to Baseline visit
* History of known hypersensitivity to any of the ingredients in APG777, APG990, or dupilumab.
* Presence of dermatologic conditions and/or comorbidities that might confound the diagnosis of AD and/or might interfere with study assessments

Note: Additional protocol defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 24 weeks

SECONDARY OUTCOMES:
Predose Serum Concentrations (Ctrough) of APG777 | Baseline, Week 1, 2, 4, 8, 12, 16, 20, 24
  PK parameters will be performed using a non-compartmental approach with a validated PK software.
Predose Serum Concentrations (Ctrough) of APG990 | Baseline, Week 1, 2, 4, 8, 12, 16, 20, 24
  PK parameters will be performed using a non-compartmental approach with a validated PK software.
Maximum Serum Concentrations (Cmax) of APG777 | Baseline, Week 1, 2, 4, 8, 12, 16, 20, 24
  PK parameters will be performed using a non-compartmental approach with a validated PK software
Maximum Serum Concentrations (Cmax) of APG990 | Baseline, Week 1, 2, 4, 8, 12, 16, 20, 24
  PK parameters will be performed using a non-compartmental approach with a validated PK software.
Time to Reach Cmax (tmax) of APG777 | Baseline, Week 1, 2, 4, 8, 12, 16, 20, 24
  PK parameters will be performed using a non-compartmental approach with a validated PK software. If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value.
Time to Reach Cmax (tmax) of APG990 | Baseline, Week 1, 2, 4, 8, 12, 16, 20, 24
  PK parameters will be performed using a non-compartmental approach with a validated PK software. If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value.

CONTACTS AND LOCATIONS:
Locations (18):
- Australia (9):
  - Investigational Site, Darlinghurst, New South Wales
  - Investigational Site, Kogarah, New South Wales
  - Investigational Site, Westmead, New South Wales
  - Investigational Site, Woolloongabba, Queensland
  - Investigational Site, Carlton, Victoria
  - Investigational Site, East Melbourne, Victoria
  - Investigational Site, Mitcham, Victoria
  - Investigational Site, Parkville, Victoria
  - Investigational Site, Fremantle, Western Australia
- Canada (7):
  - Investigational Site, London, Ontario
  - Investigational Site, Peterborough, Ontario
  - Investigational Site, Richmond Hill, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Montreal, Quebec
  - Investigational Site, Québec, Quebec
  - Investigational Site, Sherbrooke, Quebec
- New Zealand (2):
  - Investigational Site, Hamilton, Waitako
  - Investigational Site, Auckland

IPD SHARING:
Plan to Share IPD: No